CLINICAL TRIAL: NCT03258346
Title: Reversing Muscle Loss With Exercise Training and Daily Consumption of Pomegranate Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: POM Wonderful LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-05-0092
Record Dates: First submitted 2017-07-12; First posted 2017-08-23 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Sarcopenia; Cardiovascular Risk Factor
Keywords: Pomegranate Juice; Functional Tasks of Living
MeSH Terms: conditions — Sarcopenia | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Pomegranate juice will be administered in double blind placebo controlled method. Coding will be established by POM Wonderful, LLC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Pomegranate Juice (Experimental): Exercise training with daily consumption of pomegranate juice containing polyphenols
  Interventions: Other: Inertial Load Cycling Training; Dietary Supplement: Pomegranate Juice
- Exercise and Placebo (Placebo Comparator): Exercise training with daily consumption of pomegranate juice with polyphenols removed
  Interventions: Other: Inertial Load Cycling Training; Dietary Supplement: Placebo

INTERVENTIONS:
Other: Inertial Load Cycling Training — Each session of training will require a total of 15 min with the total time actually exercising of only 60-120 sec. The first week will consist of performing 15 'sprints' on the ILE, beginning each sprint with 56 sec of rest. During week 2-5, subjects will rest 41 sec between sprints, completing 20 bouts. Finally, during weeks 6-10, subjects will take 26 s rest between sprints and complete 30 bouts).
  Other Names: High intensity interval training
Dietary Supplement: Pomegranate Juice — Subjects will consume 8oz of pomegranate juice daily for duration of study.
  Arms: Exercise and Pomegranate Juice
Dietary Supplement: Placebo — Subjects will consume 8oz of pomegranate juice daily, that has had the polyphenols removed.
  Arms: Exercise and Placebo

SUMMARY:
A research study regarding the body's response to several weeks of training using short sprints and pomegranate juice supplementation

DETAILED DESCRIPTION:
The investigators have shown that chronic pomegranate juice consumption in both young untrained and weight-trained men partially protects muscles against the damage done from performing high intensity eccentric contractions and that it accelerates recovery of function. Clearly, skeletal muscle is a target for some of the healthful molecules in pomegranate juice. However, the most widespread and serious ailment to strike skeletal muscle is sarcopenia (e.g.; loss of muscle mass and becoming 'frail') with age due predominantly to a loss of 'fast-twitch' muscle fibers. Since adults rarely sprint or exert maximal force or power, they rarely use their fast-twitch muscle fibers, which thus degenerate greatly with age. Usually, about one-half of a person's muscle fibers are fast-twitch. It is the investigators' hypothesis that the combination of power exercise training and pomegranate juice supplementation (POM) over 10 weeks, will elicit greater improvements in maximal muscular power and functional physical abilities compared to power training with a placebo. The investigators also will identify changes in size and composition of leg muscles (MRI) and of the whole body (DEXA). The investigators simple logic is that muscles deteriorate with age because they are 'turned-off' and that exercise training can turn them 'back-on', but in order for the muscle fibers to fully repair when turned 'back-on' with exercise, they might benefit from agents known to foster repair, such as the natural polyphenols in pomegranate juice. It has recently been found that polyphenols are metabolized into urolithins which improve muscle cell function due to increased mitophagy. The investigators aim to determine if power training and pomegranate juice have additive effects in promoting improvements of muscle function and mass in men and women age 50-70 y.

A second purpose is to include a cardio-metabolic exercise training stimulus into the workout without compromising the efficacy of the power training. One feature of cardio-metabolic training is an increase in muscle mitochondria and oxygen utilization which might improve muscle fiber repair. The 'power training' will consist of maximal effort 4 sec sprints on a cycle ergometer with no added resistance with the only load being that of the inertia of the flywheel as the subject accelerates from 0 to their maximal RPM's while cycling (100-150 RPM)('inertial load ergometer'; ILE). The power training will be accomplished by having the subject complete 15-30 sprints in a 15 min period. During the training bouts, initially the subjects will rest 56 s between sprints (week 1- complete 15 sprints in each15 min bout), and then 41 s between sprints (weeks 2-5 and complete 20 sprints) and finally 26 s between sprints (weeks 6-10 and complete 30 sprints). The shorter rest periods (41 s and 26 s) will result in incomplete recovery of the cardio-respiratory system and thus the oxygen consumption and heart rate will average 50-70% of maximal values, which is a similar intensity as jogging, but without the jarring of foot strike.

ELIGIBILITY:
Inclusion Criteria:

* 50-70 year old male and females

Exclusion Criteria:

* not currently exercising regularly
* meets criteria for MRI scanning at Imaging Research Center at UT Austin
* history of heart disease
* knee/hip joint problems
* determination by the physician monitoring pre inclusion stress test

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Change in muscle volume | Baseline to 11 weeks
  Volume of the thigh musculature as determined by MRI analysis.
Change in sarcopenia obesity | Baseline to 11 weeks
  Intermuscular adipose tissue infiltration as measured by MRI
Change in aerobic capacity | Baseline to 11 weeks
  VO2 Max on a cycle ergometer
Change in anaerobic capacity | Baseline to 11 weeks
  The percent of maximal aerobic capacity that a subject can exercise at while not building up blood lactate
Change in muscle fatigue | Baseline to 11 weeks
  Muscle aerobic stress as measured by near infrared spectroscopy
Change in body composition | Baseline to 11 weeks
  Fat and fat free regional and total mass as measured by dual x-ray absorptiometry
Change in maximal power production | Baseline to 11 weeks
  The ability to produce power as determined on the cycle ergometer and measured in watts

SECONDARY OUTCOMES:
Change in cardiovascular risk factors | Baseline to 11 weeks
  Flow mediated dilation and pulse wave velocity
Change in urolithins | Baseline, 2 hrs after consuming first pomegranate or placebo supplement
  The ability to breakdown the beneficial components of pomegranate juice into urolithins is different among individuals
Change in Microbiome | Baseline, week 10 and week 15
  The change in the gut microbiota as a result of supplementation with pomegranate juice.
Change in maximal isometric strength | Baseline to 11 weeks
  The maximal ability to push against a immovable object as measured in the thigh musculature
Change in functional tests of living | Baseline to 11 weeks
  Movement tasks specific to the daily life of the elderly
Change in isokinetic torque | Baseline to 11 weeks
  The subject will exert maximal leg extension at two speeds and the maximal torque generated will be quantified

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Coyle, PhD, Principal Investigator — UT Austin
Locations (1):
- Human Performance Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allen JR, Satiroglu R, Fico B, Tanaka H, Vardarli E, Luci JJ, Coyle EF. Inertial Load Power Cycling Training Increases Muscle Mass and Aerobic Power in Older Adults. Med Sci Sports Exerc. 2021 Jun 1;53(6):1188-1193. doi: 10.1249/MSS.0000000000002588. PMID 33433149